CLINICAL TRIAL: NCT01237548
Title: The Evaluation of the Acute Effect of Water-Pipe Smoking on the Endothelial Function and the Respiratory System
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: Narghile Endotheil RMC 284
Record Dates: First submitted 2010-11-03; First posted 2010-11-09 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: water pipe smoking; acute effect; Endothelial; healthy adults who smoke narghile
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All participants: Normal People who have smoked Water-pipe, at least once before.
  Interventions: Other: Smoking Narghile for 30 min

INTERVENTIONS:
Other: Smoking Narghile for 30 min — No Other intervention will be used

SUMMARY:
Title: The acute effect of narghile smoking on endothelial Function, and exhaled breath condensate (EBC) and pulmonary function tests in healthy volunteers.

Objectives: To evaluate the acute effect of one cession of narghile smoking on endothelial Function, airway inflammation as assessed by exhaled breath condensate (EBC) in healthy volunteers.

Design: Prospective study evaluating these parameters before and after 30 minutes of Narghile smoking. The changes in inflammatory parameters pre and post smoking will be evaluated blindly.

Sample size: 50 participants Participant selection: Adults subjects who smoke Narghile . Intervention: Each subject will undergo evaluation including a respiratory questionnaire, endothelial Function , pulmonary function tests , exhaled breath condensate (EBC) and carboxy- hemoglobin levels . All measurements will be evaluated before and after one cession of 30 minutes narghile smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Y.O.
* Have smoked Water-pipe at least once before.

Exclusion Criteria:

* Breast feeding Women.
* S/P Bacterial Or Viral infection, Last 2 weeks
* P.O. Steroids
* Water-pipe smoking, last 24 hours
* Cigarette smoking, last 6 hours
* Intensive exposure to smoke (fire), last 24 hours
* S/P Intensive Care Hospitalization, last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal People who have smoked Water-pipe, at least once before.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
PRE - Endothelial Function as assessed by EndoPAT2000 | baseline (before smoking narghile)
  as assessed by EndoPAT2000. a pulse-oxymeter that asseses the endothelial function
POST - Endothelial Function as assessed by EndoPAT2000 | after 30 minutes of smoking narghile
  as assessed by EndoPAT2000. a pulse-oxymeter that asseses the endothelial function

SECONDARY OUTCOMES:
carboxy- hemoglobin | before and immediatly after 30 min of smoking
  Blood Test
heart rate | before and immediatly after 30 min of smoking
  Heart Beats count
Visual Analog Score 1-10 (1=bad 10=good) | before and immediatly after 30 min of smoking
  Questionnaire
Respiratory Rate | before and immediatly after 30 min of smoking
Spirometry | before and immediatly after 30 min of smoking
  Koko spirometry system
Eosinophils Count | before and immediatly after 30 min of smoking
  Blood Test
Blood Pressure | before and immediatly after 30 min of smoking
  Regular Blood Pressure assesment
Exhaled Breath Condensate | before and immediatly after 30 min of smoking
  R-tubes test

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Bentur L, Hellou E, Goldbart A, Pillar G, Monovich E, Salameh M, Scherb I, Bentur Y. Laboratory and clinical acute effects of active and passive indoor group water-pipe (narghile) smoking. Chest. 2014 Apr;145(4):803-809. doi: 10.1378/chest.13-0960. PMID 24158379